CLINICAL TRIAL: NCT01349790
Title: Prospective, Open-label, Non-controlled, Multicenter, Phase III Clinical Study to Evaluate the Efficacy and Safety of Immunoglobulin Intravenous (Human) 10% (NewGam) in Primary Immune Thrombocytopenia
Brief Title: Efficacy and Safety of Immunoglobulin Intravenous (Human) 10% (NewGam) in Primary Immune Thrombocytopenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGAM-02; 2009-014589-24 (EudraCT Number)
Record Dates: First submitted 2011-05-05; First posted 2011-05-09 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: Primary Thrombocytopenia
Keywords: ITP; Primary immune thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NewGam (Experimental): Each participant received 1 g/kg NewGam intravenously on 2 consecutive days.
  Interventions: Drug: NewGam

INTERVENTIONS:
Drug: NewGam — NewGam is a solution of human normal immunoglobulin 10% treated with solvent/detergent and nanofiltered for intravenous administration.

SUMMARY:
NewGam is a newly developed human normal immunoglobulin solution for intravenous administration (IGIV). This study will evaluate the safety and efficacy of NewGam 10% in patients with primary immune thrombocytopenia.

DETAILED DESCRIPTION:
The primary objective of the study is to assess the efficacy of NewGam in correcting the platelet count. The secondary objective of the study is to evaluate the safety of NewGam. Safety will be assessed by monitoring vital signs, physical examination, evaluation of adverse events (AE) and laboratory parameters, and viral safety testing.

ELIGIBILITY:
Inclusion Criteria:

1. Age of ≥ 18 and ≤ 65 years.
2. Confirmed diagnosis of chronic primary immune thrombocytopenia (ITP) (diagnosed with a threshold platelet count < 100x10^9/L) of at least 12 months duration.
3. Platelet count of no more than 20x10^9/L with or without bleeding manifestations.
4. Freely given written informed consent from patient.
5. Women of childbearing potential must have a negative result on a pregnancy test (human chorionic gonadotropin [HCG]-based assay) and need to practice contraception using a method of proven reliability for the duration of the study.

Exclusion Criteria:

1. Thrombocytopenia secondary to other diseases (such as acquired immunodeficiency syndrome [AIDS] or systemic lupus erythematosus [SLE]), or drug-related thrombocytopenia.
2. Administration of intravenous immunoglobulin (IGIV), anti-D immunoglobulin or thrombopoietin receptor agonists, or other platelet enhancing drugs (including immunosuppressive or other immunomodulatory drugs) within 3 weeks before enrollment, except for:

   * Long-term corticosteroid therapy when the dose has been stable during the preceding 3 weeks and no dosage change is planned until study Day 22.
   * Long-term azathioprine, cyclophosphamide, or attenuated androgen therapy when the dose has been stable during the preceding 3 months and no dosage change is planned until study Day 22.
3. Unresponsive to previous treatment with IGIV or anti-D immunoglobulin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abdulgabar Salama, MD, Principal Investigator — Universitätsklinikum Charite, Med. Fakultät der Humboldt-Universität Berlin; Wolfgang Frenzel, MD, Study Director — Octapharma AG
Locations (1):
- Abdulgabar Salama, Berlin, Germany

REFERENCES:
- [Derived] Arbach O, Taumberger AB, Wietek S, Cervinek L, Salama A. Efficacy and safety of a new intravenous immunoglobulin (Panzyga(R) ) in chronic immune thrombocytopenia. Transfus Med. 2019 Feb;29(1):48-54. doi: 10.1111/tme.12573. Epub 2019 Jan 27. PMID 30687970

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NewGam
Started | 40
Completed | 31
Not Completed | 9
Not completed — Investigator Judgement | 3
Not completed — Death | 2
Not completed — Withdrawal by Patient | 2
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Safety set: All participants enrolled in the study who received at least part of 1 dose of NewGam.
Arm/Group | NewGam
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (15.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders
Description: A responder is a study participant with an increase in platelets to ≥ 50x10^9/L within 7 days after the first infusion, ie, by study Day 8.
Time Frame: Day 1 to Day 8
Population: Full analysis set: All participants enrolled in the study who received at least part of 1 dose of NewGam and who had at least 1 post-baseline measurement of platelet concentration.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NewGam
Number analyzed (Participants) | 36
Percentage of participants | 80.6 [63.98 to 91.81]

2. Secondary Outcome: Percentage of Alternative Responders
Description: An alternative responder is a study participant with an increase in platelets to ≥ 30x10^9/L and to at least double the baseline platelet count, confirmed on at least 2 occasions at least 7 days apart, and absence of bleeding.
Time Frame: Day 1 to Day 22
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NewGam
Number analyzed (Participants) | 36
Percentage of participants | 66.7 [49.03 to 81.44]

3. Secondary Outcome: Percentage of Complete Responders
Description: A complete responder is a study participant with an increase in platelets to ≥ 100x10^9/L, confirmed on at least 2 occasions at least 7 days apart, and absence of bleeding.
Time Frame: Day 1 to Day 22
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NewGam
Number analyzed (Participants) | 36
Percentage of participants | 50.0 [32.92 to 67.08]

4. Secondary Outcome: Percentage of Alternative Responders Who Lost the Response
Description: An alternative responder who lost the response is a study participant who met the criterion for an alternative response but who then deteriorated, ie, their platelet count decreased to < 30x10^9/L, their platelet count decreased to less than double the baseline count, or bleeding occurred.
Time Frame: Day 1 to Day 22
Population: Full analysis set: All participants enrolled in the study who received at least part of 1 dose of NewGam and who had at least 1 post-baseline measurement of platelet concentration. Only participants with an alternative response were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NewGam
Number analyzed (Participants) | 24
Percentage of participants | 45.8 [25.55 to 67.18]

5. Secondary Outcome: Percentage of Complete Responders Who Lost the Response
Description: A complete responder who lost the response is a study participant who met the criterion for a complete response but who then deteriorated, ie, their platelet count decreased to < 100x10^9/L or bleeding occurred.
Time Frame: Day 1 to Day 22
Population: Full analysis set: All participants enrolled in the study who received at least part of 1 dose of NewGam and who had at least 1 post-baseline measurement of platelet concentration. Only participants with a complete response were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NewGam
Number analyzed (Participants) | 18
Percentage of participants | 77.8 [52.36 to 93.49]

6. Secondary Outcome: Time to a Response
Description: A study participant had a response if their platelets increased to ≥ 50x10^9/L within 7 days after the first infusion, ie, by study Day 8.
Time Frame: Day 1 to Day 8
Population: Full analysis set: All participants enrolled in the study who received at least part of 1 dose of NewGam who had at least 1 post-baseline measurement of platelet concentration. Only responders were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | NewGam
Number analyzed (Participants) | 29
Days | 2.0 [1.00 to 2.00]

7. Secondary Outcome: Time to an Alternative Response
Description: A study participant had a response if their platelets increased to ≥ 30x10^9/L and to at least double the baseline platelet count, confirmed on at least 2 occasions at least 7 days apart, and absence of bleeding.
Time Frame: Day 1 to Day 22
Population: Full analysis set: All participants enrolled in the study who received at least part of 1 dose of NewGam who had at least 1 post-baseline measurement of platelet concentration. Only participants with an alternative response were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | NewGam
Number analyzed (Participants) | 24
Days | 1.0 [1.00 to 2.00]

8. Secondary Outcome: Time to a Complete Response
Description: A study participant had a complete response if their platelets increased to ≥ 100x10^9/L, confirmed on at least 2 occasions at least 7 days apart, and absence of bleeding.
Time Frame: Day 1 to Day 22
Population: Full analysis set: All participants enrolled in the study who received at least part of 1 dose of NewGam who had at least 1 post-baseline measurement of platelet concentration. Only participants with a complete response were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | NewGam
Number analyzed (Participants) | 18
Days | 2.0 [2.00 to 2.00]

9. Secondary Outcome: Duration of a Response
Description: The duration of a response was defined as the time from when a response was achieved until the platelet count fell below 50x10^9/L.
Time Frame: Day 1 to Day 22
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | NewGam
Number analyzed (Participants) | 29
Days | 14.0 [10.00 to 17.00]

10. Secondary Outcome: Duration of an Alternative Response
Description: The duration of an alternative response was defined as the time from when an alternative response was achieved until the platelet count fell below 50x10^9/L.
Time Frame: Day 1 to Day 22
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | NewGam
Number analyzed (Participants) | 24
Days | 18.5 [17.00 to 20.00]

11. Secondary Outcome: Duration of a Complete Response
Description: The duration of a complete response was defined as the time from when a complete response was achieved until the platelet count fell below 50x10^9/L.
Time Frame: Day 1 to Day 22
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | NewGam
Number analyzed (Participants) | 18
Days | 12.5 [10.00 to 16.00]

12. Secondary Outcome: Platelet Count by Visit
Description: The platelet count at each study visit are presented.
Time Frame: Day 1 to Day 22
Population: Full analysis set: All participants enrolled in the study who received at least part of 1 dose of NewGam who had at least 1 post-baseline measurement of platelet concentration.
Measure: Mean (Standard Deviation); unit: 10^9 platelets/L
Arm/Group | NewGam
Number analyzed (Participants) | 36
10^9 platelets/L
  Baseline | 8.8 (5.76)
  Day 2 | 41.6 (31.41)
  Day 3 | 115.0 (85.58)
  Day 4 | 154.6 (118.04)
  Day 5 | 168.2 (149.89)
  Day 6 | 179.3 (178.64)
  Day 7 | 206.3 (195.75)
  Day 8 | 186.5 (205.44)
  Day 15 | 88.1 (130.07)
  Day 22/End of treatment | 41.4 (65.48)

13. Secondary Outcome: Maximum Platelet Count
Description: The maximum platelet count achieved during the study is presented.
Time Frame: Day 1 to Day 22
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: 10^9 platelets/L
Arm/Group | NewGam
Number analyzed (Participants) | 36
10^9 platelets/L | 236.9 (205.18)

14. Secondary Outcome: Percentage of Responders Who Achieved a Normal Platelet Count
Description: The percentage of responders who achieved a normal platelet count is presented.
Time Frame: Day 1 to Day 22
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NewGam
Number analyzed (Participants) | 29
Percentage of participants | 79.3 [60.28 to 92.01]

15. Secondary Outcome: Bleeding Intensity
Description: The percentage of participants with various intensities of overall bleeding, epistaxis (bleeding of the nose), oral bleeding, and skin bleeding graded as none, minor, mild, moderate, or severe at Baseline and Day 22 are reported.
Time Frame: Day 1 to Day 22
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | NewGam
Number analyzed (Participants) | 36
Percentage of participants
  Overall - Total - Baseline | 100.0
  Overall - Total - Day 8 | 100.0
  Overall - Total - Day 22 | 100.0
  Overall - None - Baseline | 36.1
  Overall - None - Day 8 | 91.2
  Overall - None - Day 22 | 72.2
  Overall - Minor - Baseline | 38.9
  Overall - Minor - Day 8 | 5.9
  Overall - Minor - Day 22 | 19.4
  Overall - Mild - Baseline | 5.6
  Overall - Mild - Day 8 | 2.9
  Overall - Mild - Day 22 | 2.8
  Overall - Moderate - Baseline | 19.4
  Overall - Moderate - Day 8 | 0.0
  Overall - Moderate - Day 22 | 2.8
  Overall - Severe - Baseline | 0.0
  Overall - Severe - Day 8 | 0
  Overall - Severe - Day 22 | 2.8
  Epistaxis - Total - Baseline | 100.0
  Epistaxis - Total - Day 22 | 100.0
  Epistaxis - None - Baseline | 83.3
  Epistaxis - None - Day 22 | 91.7
  Epistaxis - Minor - Baseline | 8.3
  Epistaxis - Minor - Day 22 | 8.3
  Epistaxis - Mild - Baseline | 5.6
  Epistaxis - Mild - Day 22 | 0.0
  Epistaxis - Moderate - Baseline | 2.8
  Epistaxis - Moderate - Day 22 | 0.0
  Epistaxis - Severe - Baseline | 0.0
  Epistaxis - Severe - Day 22 | 0.0
  Oral bleeding - Total - Baseline | 100.0
  Oral bleeding - Total - Day 22 | 100.0
  Oral bleeding - None - Baseline | 75.0
  Oral bleeding - None - Day 22 | 86.1
  Oral bleeding - Minor - Baseline | 13.9
  Oral bleeding - Minor - Day 22 | 8.3
  Oral bleeding - Mild - Baseline | 0.0
  Oral bleeding - Mild - Day 22 | 2.8
  Oral bleeding - Moderate - Baseline | 5.6
  Oral bleeding - Moderate - Day 22 | 2.8
  Oral bleeding - Severe - Baseline | 5.6
  Oral bleeding - Severe - Day 22 | 0.0
  Skin bleeding - Total - Baseline | 100.0
  Skin bleeding - Total - Day 22 | 100.0
  Skin bleeding - None - Baseline | 41.7
  Skin bleeding - None - Day 22 | 77.8
  Skin bleeding - Minor - Baseline | 25.0
  Skin bleeding - Minor - Day 22 | 22.2
  Skin bleeding - Mild - Baseline | 27.8
  Skin bleeding - Mild - Day 22 | 0.0
  Skin bleeding - Moderate - Baseline | 5.6
  Skin bleeding - Moderate - Day 22 | 0.0
  Skin bleeding - Severe - Baseline | 0.0
  Skin bleeding - Severe - Day 22 | 0.0

16. Secondary Outcome: Percentage of Participants Who Achieved a Platelet Count > 30x10^9/L
Description: The percentage of participants who achieved a platelet count > 30x10^9/L within 1 and 2 days after infusion is reported.
Time Frame: Day 1 to Day 2
Population: Safety set: All participants enrolled in the study who received at least part of 1 dose of NewGam.
Measure: Number; unit: Percentage of participants
Arm/Group | NewGam
Number analyzed (Participants) | 40
Percentage of participants
  Day 1 | 55.0
  Day 2 | 77.5

ADVERSE EVENTS:
Description: Safety set: All participants enrolled in the study who received at least part of 1 dose of NewGam.
Arm/Group | NewGam
Serious Adverse Events (participants affected / at risk) | 6/40
Other Adverse Events (participants affected / at risk) | 30/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NewGam (N=40)
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Cerebral haematoma (Nervous system disorders) | 1
Meningitis aseptic (Nervous system disorders) | 1
Pneumonia (Infections and infestations) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NewGam (N=40)
Headache (Nervous system disorders) | 17
Dizziness (Nervous system disorders) | 3
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 6
Anaemia (Blood and lymphatic system disorders) | 5
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 2
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 2
Chills (General disorders) | 2
Pyrexia (General disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No